CLINICAL TRIAL: NCT04258254
Title: A Multisystem, Multimodal Intervention for Children With ASD
Brief Title: The Effect of Play on Social and Motor Skills of Children With ASD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1539736-1; 3P20GM103446-19S1 (NIH)
Record Dates: First submitted 2020-01-24; First posted 2020-02-06 (Actual); Results first posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Movement; Play; Social; Communication; Motor
MeSH Terms: conditions — Autism Spectrum Disorder; Communication | interventions — Combined Modality Therapy; Exercise; Standard of Care

STUDY DESIGN:
Intervention Model Description: Participating children are matched on age, gender, and level of functioning. Matched pairs will be randomized to a) multimodal or b) general movement or c) standard of care, seated play group.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Multimodal (Experimental): Each child will receive 16 training sessions (8 weeks of training @ 2 sessions per week, approximately 30-45 minutes of interaction time per session) from an expert trainer and parent guidance using telehealth or face-to-face interactions. Within each session, the child will engage in tasks requiring interpersonal synchrony, multilimb coordination (asymmetrical and ipsi/contralateral motions), and balance. Based on feasibility, parents will be given appropriate supplies and trained to promote similar activities at home 1-2 days/week.
  Interventions: Behavioral: Multimodal
- General Movement (Active Comparator): Each child will receive 16 training sessions (8 weeks of training @ 2 sessions per week, approximately 30-45 minutes of interaction time per session) from an expert trainer and parent guidance using telehealth or face-to-face interactions. Within each session, the child will engage in structured physical activity focused on flexibility, strength, and endurance. Based on feasibility, parents will be given appropriate supplies and trained to promote similar activities at home 1-2 days/week.
  Interventions: Behavioral: General
- Standard of Care (Active Comparator): Each child will receive 16 training sessions (8 weeks of training @ 2 sessions per week, approximately 30-45 minutes of interaction time per session) from an expert trainer and parent guidance using telehealth or face-to-face interactions. Within each session, the child will engage in seated play focused on reading, building, and art-craft activities. Based on feasibility, parents will be given appropriate supplies and trained to promote similar activities at home 1-2 days/week.
  Interventions: Behavioral: Standard of Care

INTERVENTIONS:
Behavioral: Multimodal — Multimodal intervention will involve hello songs, warm up mainly involve sensory and stretching games, music time involves playing instruments, moving game involves use of music or songs to move the whole body, yoga involves themes/songs to perform yoga poses, and good bye involves a goodbye song and reflections about the session. In all movement conditions, trainers emphasize complex and multilimb coordination (asymmetrical and ipsi/contralateral movements) and balance.
  Other Names: Coordination/Balance
  Arms: Multimodal
Behavioral: General — The general exercise group will begin with hello games/set up and end with reflections and cleanup. Children will engage in limb and body warmup routines, specific strengthening exercises (single-joint/single-limb/symmetrical), moderate intensity endurance exercises involving various obstacle courses, and a cool down routine.
  Other Names: Physical Activity, Strength, Endurance
  Arms: General Movement
Behavioral: Standard of Care — The seated play group will also begin with hello/icebreaker games and end with goodbye and cleanup. In between, they will read books and review the story line and overall message and engage in fine-motor activities involving building supplies and art-craft.
  Other Names: Sedentary or Seated Play
  Arms: Standard of Care

SUMMARY:
In this study, the investigators will compare effects of two types of 8-weeklong interventions: a) multimodal or b) general movement to facilitate social communication and motor skills of school-age children with Autism Spectrum Disorder (ASD). Recently, the investigators have identified cortical dysfunction patterns as markers of imitation/interpersonal synchrony difficulties in children with ASD using functional near-infrared spectroscopy. In this project, the investigators want to validate whether cortical markers can determine treatment responders and if such markers are sensitive to training-related changes. Following training, the investigators expect to see a variety of behavioral and neural changes in both groups. If the study aims are achieved, the investigators will validate the use of cortical markers as a treatment response measure. This research will build evidence for the use of various movement interventions for school-age children with ASD.

DETAILED DESCRIPTION:
46 children with ASD between 5 and 15 years of age will be randomly assigned to the multimodal or general play or seated play groups. Each child will participate in 9 testing sessions (4 pretests, 3 posttests, and 3, 2-month follow-ups) and 8 weeks of multimodal or general intervention between pre-tests and post-tests. In the 8-week phase between the pre- and post-tests, each child will complete group-specific intervention-related activities with the expert clinician twice per week via telehealth or face-to-face interactions. Each session will last for around 1-1.5 hours. If the study aims are achieved, the investigators will validate the use of cortical markers as a treatment response measure. Findings from this research will offer evidence for the use of various movement interventions to promote motor, social communication, and cognitive skills in school-age children with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Children with Autism Spectrum Disorder (ASD) between 5 and 15 years of age

Exclusion Criteria:

* Significant hearing or vision impairment
* Significant behavioral problems
* Significant medical (cardiovascular or respiratory), orthopedic, or surgical problems that prevent study participation.
* History of seizures.
* Significant mobility problems that prevent study participation.

Ages: 5 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 46 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anjana N Bhat, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Su WC, Cleffi C, Srinivasan S, Bhat A. A Pilot Study Comparing the Efficacy, Fidelity, Acceptability, and Feasibility of Telehealth and Face-to-Face Creative Movement Interventions in Children with Autism Spectrum Disorder. Telemed Rep. 2024 Mar 21;5(1):67-77. doi: 10.1089/tmr.2023.0061. eCollection 2024. PMID 38558955

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multimodal | General Movement | Standard of Care
Started | 15 | 16 | 15
Completed | 15 | 15 | 15
Not Completed | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multimodal | General Movement | Standard of Care | Total
Number analyzed (Participants) | 15 | 16 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (0.6) | 9.1 (0.6) | 8.4 (0.6) | 9 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 4 | 2 | 9
  Male | 12 | 12 | 13 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 10 | 7 | 8 | 25
  African American | 3 | 2 | 5 | 10
  Asian | 2 | 7 | 2 | 11
Vineland Adaptive Behavior Scales, ABC Score [Mean (Standard Deviation); unit: units on a scale] | 71.4 (3) | 70.4 (2.9) | 75.5 (2.8) | 72 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2)
Description: The 3 gross motor coordination and 1 fine manual control composite of the Bruininks-Oseretsky Test of Motor Proficiency-Second Edition (BOT-2) were administered as a measure of gross and fine motor coordination at each time point. BOT-2 standard scores will be reported for each composite: (i) body coordination composite comprises of balance and bilateral coordination, (ii) the strength/agility composite is comprised of running speed and agility, (iii) upper-limb coordination composite is comprised of upper-limb coordination and manual dexterity, and (iv) the fine manual control composite is comprised of fine motor precision and integration. Standard composite scores on the BOT-2 have a Mean=50 and a standard deviation (SD)=10 for body coordination, strength & agility, manual coordination and fine motor coordination composite domains. Higher standard scores represent a better outcome. Note there are no T-scores as such for BOT-2; the term often used is a standard BOT composite score.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Population: Standard composite scores (Mean=50, SD=10) for body coordination, strength & agility, manual coordination and fine motor coordination.
Measure: Mean (Standard Error); unit: score on a scale BOT-2
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
score on a scale BOT-2
  Pretest BOT body coordination | 36.4 (2.0) | 36.9 (3.6) | 36.5 (1.9)
  Posttest BOT Body Coordination | 40.9 (2.8) | 44.0 (3.8) | 37.7 (1.9)
  Follow-up BOT Body coordination | 40.8 (2.5) | 44 (3.7) | 37 (1.8)
  Pretest BOT Strength&Agility | 32.3 (2.2) | 37.4 (2.9) | 33.3 (1.6)
  Posttest BOT Strength & Agility | 34.5 (2.7) | 42.5 (3.0) | 34.4 (1.9)
  Follow-up BOT Strength & Agility | 33 (2.3) | 43 (3.1) | 33.4 (1.7)
  Pretest BOT Manual Coordination | 29.8 (1.4) | 33.3 (1.5) | 33.0 (1.5)
  Posttest BOT Manual Coordination | 31.1 (2.3) | 34.5 (1.4) | 33.3 (1.6)
  Follow-Up BOT Manual Dexterity | 32 (2.0) | 33 (1.2) | 34 (1.7)
  Pretest BOT Fine-manual control | 36.4 (2.7) | 40.7 (3.1) | 36.4 (2.4)
  Posttest BOT Fine manual control | 36.1 (2.8) | 41.4 (3.4) | 41.5 (2.5)
  Follow-up BOT Fine manual control | 37 (2.5) | 41 (2.9) | 42.3 (2.2)

2. Primary Outcome: Praxis Subtests of the Sensory Integration and Praxis Testing (SIPT) - Postural Praxis Error
Description: The praxis subtests of Sensory Integration and Praxis Testing (SIPT) are standardized and normed measures of examining motor coordination, sensory integration, and praxis. Specifically, the investigators are planning to use items from subtest of postural praxis subtest. The praxis subtests will examine a child's ability to generalize the imitation skills to novel actions involved in the SIPT postural praxis subtest. This test provides the number of errors per action copied and a total number of errors. There is no fixed range as such but the scores could range from 0 to 100. There are no T or standard scores available for this subtest. Higher number of errors indicates a poor outcome.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Measure: Mean (Standard Error); unit: number of errors
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
number of errors
  Pretest Total Praxis Error | 21.5 (1.5) | 23.1 (1.8) | 22.4 (2.0)
  Posttest Total Praxis Error | 17.6 (1.5) | 20.1 (1.6) | 17 (2.2)
  Follow-Up Total Praxis Error | 15.9 (2.3) | 18.7 (1.9) | 18.1 (1.6)

3. Primary Outcome: Flanker Task of Executive Functioning (EF)
Description: In the EF task data will be collected. Children will completed the response inhibition task using the Flanker test. This involves making decisions about where a group of fish shown on the screen are looking (right or left). Reaction time in msec were calculated for each response and averaged across trials. Lower values of reaction times indicate faster or better responses.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Measure: Mean (Standard Error); unit: Reaction time in msec
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 9 | 14 | 13
Reaction time in msec
  Pretest Incongruent condition, Flanker Reaction Time | 3.6 (0.9) | 2.4 (0.5) | 2.1 (0.5)
  Posttest Incongruent condition, Flanker Reaction Time | 2.4 (0.65) | 1.8 (0.6) | 1.9 (0.6)
  Followup Incongruent Flanker Reaction Time | 2.4 (0.6) | 2.0 (0.6) | 1.9 (0.5)

4. Primary Outcome: Synchrony Errors During the Rhythmic Synchrony Task
Description: In the rhythmic synchrony task children will perform social drumming (i.e., move in synchrony with an adult as the child follows the adult's drumming motions). Synchrony errors were coded when the child was not matching with the adult for each movement cycle. Higher number of errors indicate a poor outcome. This was an experimental paradigm, and not a standardize measure. Hence, there are no T-scores to report.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Population: Number of errors.
Measure: Mean (Standard Error); unit: Number of erroneous cycles
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
Number of erroneous cycles
  Pretest Social Synchrony error # | 1.9 (0.1) | 1.9 (0.2) | 2.1 (1.3)
  Posttest Social Synchrony error # | 1.3 (0.2) | 1.4 (0.2) | 2 (0.1)
  Follow-up Social Synchrony error # | 1.5 (0.2) | 1.6 (0.2) | 1.7 (0.2)

5. Primary Outcome: Number of Prosocial Behaviors
Description: In a structured play task, the tester assessed a child's ability to engage in prosocial behaviors across multiple helping bids to engage the child in helping behaviors (e.g., clean up of pennies, peg, blocks, cards, and dropped pencils). There are no T or standard scores available for this behavioral measure (not a standardized test). Higher number indicates more prosocial behaviors by the child during the helping bids.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Measure: Mean (Standard Error); unit: Number of prosocial behaviors
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
Number of prosocial behaviors
  Pretest Prosocial Behaviors # | 8.4 (0.37) | 9.3 (0.3) | 7.4 (0.8)
  Posttest Prosocial Behaviors # | 9 (0.37) | 8.6 (0.4) | 8.9 (0.4)
  Follow-up Prosocial Behaviors # | 8.8 (0.4) | 8.3 (0.6) | 7.9 (0.5)

6. Secondary Outcome: 2-Minute Walk Test
Description: Testers will use the 2-minute walk test to assess endurance of the participating children. The test will be chosen based on the walking tolerance of the child and the severity of locomotor impairments. The test assesses the maximum distance that the child can cover in 1 or 2 minutes. The 2-minute walk test distance has been found to be highly correlated with the gold standard 6-minute walk test commonly used to assess endurance. This test provides a distance measure and more the distance covered indicates better performance. The distance covered may range from 125-200 meters approximately. There are no T or standard scores available for this functional measure. Higher distance covered number indicates a better outcome.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Measure: Mean (Standard Error); unit: distance covered in feet
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 14 | 14 | 14
distance covered in feet
  Pretest 2MWT distance | 481.9 (57.8) | 416 (37.6) | 471.3 (26.9)
  Posttest 2MWT distance | 496.9 (40.2) | 478.9 (34.8) | 497.1 (24.1)
  Follow-up 2MWT distance | 405.9 (23.6) | 469.4 (38.9) | 449.4 (37)

7. Secondary Outcome: Timed-Up & Go Test (TUG)
Description: The Timed-Up & Go test (TUG) measures the time taken in seconds to stand up from a chair with armrest, walk 3 meters, turn around, walk back to the chair, and sit down again. A higher value indicates poor performance and time taken is usually between 4 to 7 seconds. There are no T or standard scores available for this functional measure. Lower value of time taken indicates better outcome.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Measure: Mean (Standard Error); unit: Time taken in seconds
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 14 | 14 | 14
Time taken in seconds
  Pretest TUG score | 7.1 (0.6) | 6.3 (0.5) | 7.3 (0.5)
  Posttest TUG score | 6.1 (0.4) | 6.3 (0.4) | 7.3 (0.5)
  Follow-up TUG score | 6.2 (0.3) | 5.5 (0.3) | 6.6 (0.4)

8. Secondary Outcome: Developmental Coordination Disorder-Questionnaire
Description: Motor coordination questionnaire provides a total score of motor performance. For Children Ages 5 years 0 months to 7 years 11 months, a score between 15 to 46 is an indication of DCD or suspect DCD and a score between 47 to 75 is probably not DCD.
  For Children Ages 8 years 0 months to 9 years 11 months, a score of 15 to 55 is an indication of DCD or suspect DCD and a score between 56 to 75 is probably not DCD.
  For Children Ages 10 years 0 months to 15 years, a score of 15 to 57 is an indication of DCD or suspect DCD and a score between 58 to 75 is probably not DCD.
  Higher number indicates better motor performance. There are no other T-scores associated with this measure.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
score on a scale
  Pretest Total DCD-Q score | 41.3 (2.7) | 44.3 (2.6) | 41.2 (1.9)
  Posttest Total DCD-Q score | 42.9 (2.7) | 48.9 (2.6) | 44.3 (1.8)
  Follow-up Total DCD-Q score | 42.8 (2.3) | 47.8 (3.1) | 44.1 (1.9)

9. Secondary Outcome: Sensory Processing Measure (SPM)
Description: Sensory Processing Measure (SPM) measures assesses challenges with social participation as well as sensory challenges. A standard T-score of 60-70 indicates some problems and a range of 70-80 indicates definite problems. Note the SPM T-score has a mean of 50 and a standard deviation (SD) of 10. Note a higher T-score indicates greater sensory processing problems.
Time Frame: Baseline to Post-test after 8 weeks of intervention, Baseline to Follow-up testing after 8 weeks from post-test
Population: T score
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 14 | 14 | 14
score on a scale
  Pretest SPM T score | 67.4 (1.7) | 68.9 (1.4) | 65 (1.6)
  Post-test SPM T score | 66.9 (1.9) | 66.3 (1.4) | 64.9 (1.7)
  Follow-up test SPM T score | 67 (1.8) | 65.9 (1.3) | 64.5 (1.9)

10. Other Pre Specified Outcome: Social Communication Questionnaire (SCQ)
Description: The Social Communication Questionnaire (SCQ) is a 15-minute parent questionnaire to screen for autism-specific, social communication behaviors of children above three years of age. A higher SCQ total score indicates a greater social communication delay. The SCQ scores may range from 0 to 39. There are no T or standard scores available for this screening measure. Higher number indicates more autistic severity.
Time Frame: In the screening phase after initial contact with researchers
Measure: Mean (Standard Error); unit: Total score
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 15 | 15 | 15
Total score | 18 (1.8) | 13 (1.5) | 13.1 (1)

11. Other Pre Specified Outcome: Vineland Adaptive Behavioral Scales (VABS)
Description: The Vineland Adaptive Behavioral Scales (VABS) is a 20-minute parent questionnaire/interview that assess a child's overall development/adaptive functioning and includes subscales of motor (gross motor, fine motor), socialization (interpersonal relationships, play, and coping skills), and communication (receptive, expressive, and written language) as well as adaptive functioning (personal, domestic, and community) for individuals between birth to 90 years of age. The VABS will provides us information on overall functioning based on the adaptive behavior composite (ABC) score. All participants will complete this measure to receive an ABC score of overall functioning. A higher VABS standard score indicates better functional performance for a given subdomain or overall. The VABS standard scores range from 1-100 with 100 being best performance.
Time Frame: In the baseline period
Measure: Mean (Standard Error); unit: Standard score
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 14 | 14 | 14
Standard score | 71 (2.9) | 77.1 (2.9) | 75.5 (2.9)

12. Other Pre Specified Outcome: Social Responsiveness Scale-Second Edition (SRS-2)
Description: Social Responsiveness Scale-Second Edition (SRS-2)(Constantino, 2012) (10 minutes): The SRS is a survey instrument designed to measure autism severity (i.e., social skill deficits that are commonly experienced by individuals with autism spectrum disorders). The SRS includes survey questions that measure skills across five different domains: Social Awareness, Social Cognition, Social Communication, Social Motivation, and Restricted Interests and Repetitive Behavior. An overall T-score of <59 is within the normal range, 60-75 is a mild-to-moderate impairment, and a T-score >75 indicates a severe impairment. Note the SRS T-score has a mean of 50 and a standard deviation (SD) of 10. Note a higher T-score indicates greater autistic severity.
Time Frame: Only completed once at pretest.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Multimodal | General Movement | Standard of Care
Number analyzed (Participants) | 14 | 14 | 14
score on a scale | 78 (2.9) | 70 (2) | 74.1 (1.5)

ADVERSE EVENTS:
Time Frame: 1 year, 6 months
Description: There is no difference in how we define adverse events.
Arm/Group | Multimodal | General Movement | Standard of Care
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/16 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/16 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04258254/Prot_002.pdf
  • Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/54/NCT04258254/SAP_003.pdf
  • Informed Consent Form (2020-12-10): https://cdn.clinicaltrials.gov/large-docs/54/NCT04258254/ICF_004.pdf